CLINICAL TRIAL: NCT03924869
Title: A Phase 3, Randomized, Placebo-Controlled Clinical Study to Evaluate the Safety and Efficacy of Stereotactic Body Radiotherapy (SBRT) With or Without Pembrolizumab (MK-3475) in Participants With Unresected Stages I or II Non Small Cell Lung Cancer (NSCLC) (KEYNOTE-867)
Brief Title: Efficacy and Safety Study of Stereotactic Body Radiotherapy (SBRT) With or Without Pembrolizumab (MK-3475) in Adults With Unresected Stage I or II Non-Small Cell Lung Cancer (NSCLC) (MK-3475-867/KEYNOTE-867)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated for business reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3475-867; MK-3475-867 (Other: MSD); KEYNOTE-867 (Other: MSD); 194909 (Registry Identifier: JAPAC-CTI); 2022-500413-11-00 (Registry Identifier: EU CT); U1111-1275-8515 (Registry Identifier: UTN); 2018-004320-11 (EudraCT Number)
Record Dates: First submitted 2019-04-22; First posted 2019-04-23 (Actual); Results first posted 2025-05-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Programmed Cell Death Receptor Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — Radiosurgery; pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SBRT + Pembrolizumab (Experimental): Participants receive SBRT once every 3 days for 3, 4, 5, or 8 fractions (dependent on tumor type/location; 45-70 Gray [Gy] total) over approximately 2 weeks PLUS pembrolizumab 200 mg via intravenous (IV) infusion once every 3 weeks for up to 17 cycles (up to approximately 1 year). Each cycle is 21 days.
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT); Biological: Pembrolizumab
- SBRT + Placebo (Placebo Comparator): Participants receive SBRT once every 3 days for 3, 4, 5, or 8 fractions (dependent on tumor type/location; 45-70 Gy total) over approximately 2 weeks PLUS placebo (normal saline solution) via IV infusion once every 3 weeks for up to 17 cycles (up to approximately 1 year). Each cycle is 21 days.
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT); Drug: Placebo

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy (SBRT) — SBRT will be administered once every 3 days for 3, 4, 5, or 8 fractions (dependent on tumor type/location; 45-70 Gray [Gy] total) over approximately 2 weeks.
Biological: Pembrolizumab — Pembrolizumab will be administered at 200 mg via IV infusion once every 3 weeks for up to 17 cycles (up to approximately 1 year).
  Other Names: MK-3475; KEYTRUDA®
  Arms: SBRT + Pembrolizumab
Drug: Placebo — Placebo (normal saline solution) will be administered at 200 mg via IV infusion once every 3 weeks for up to 17 cycles (up to approximately 1 year).
  Arms: SBRT + Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of stereotactic body radiotherapy (SBRT) plus pembrolizumab (MK-3475) in the treatment of adult participants with unresected Stage I or II (Stage IIB N0, M0) non-small cell lung cancer (NSCLC).

The primary study hypothesis is SBRT plus pembrolizumab prolongs Event-free Survival (EFS) compared to SBRT plus placebo (normal saline solution).

DETAILED DESCRIPTION:
As of protocol amendment 8, the study was stopped due to an interim analysis that did not support the study primary and key secondary endpoints. All study participants stopped ongoing treatment with pembrolizumab/placebo, and must complete end of trial and safety follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Has previously untreated non-small cell lung cancer (NSCLC) diagnosed by histology or cytology and confirmed as Stage I or II (T1 to limited T3, N0, M0) NSCLC (American Joint Committee on Cancer, AJCC) by chest computed tomography (CT) and positron emission tomography (PET) scan. Participants with pericardium invasion, >2 nodules or 2 nodules that cannot be treated in one field (>2 cm apart and/or total planned target volume [PTV] >163 cc) and diaphragm elevation suggestive of phrenic nerve invasion are excluded
* Cannot undergo thoracic surgery due to existing medical illness(es) as determined by the site's multi-disciplinary tumor board. Medically operable participants who decide to treat with stereotactic body radiotherapy (SBRT) as definitive therapy rather than surgery are also eligible, if patient's unwillingness to undergo surgical resection is clearly documented
* Has a Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
* Is able to receive SBRT and does not have an ultra-centrally located tumor
* Has adequate organ function within 7 days prior to the start of study treatment
* A female is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: a) not a women of childbearing potential (WOCBP) OR b) A WOCBP and uses contraceptive method that is highly effective (with a failure rate of <1% per year), or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis), during the intervention period and for at least 120 days after the last dose of pembrolizumab/placebo and 180 days after the last radiotherapy dose
* Male participants are eligible to participate if they agree to the following during the intervention period and for at least 90 days after the last dose of radiotherapy: refrain from donating sperm plus either be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent or must agree to use contraception per study protocol, unless confirmed to be azoospermic
* Has a radiation therapy plan approved by the central radiation therapy quality assurance vendor

Exclusion Criteria:

* Has received prior therapy with an anti-programmed cell death-1 (anti-PD-1), anti-programmed cell death-ligand 1 (anti-PD-L1), or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. cytotoxic T-lymphocyte-associated antigen 4 [CTLA-4], tumor necrosis factor receptor superfamily member 4 [OX-40], tumor necrosis factor receptor superfamily member 9 [CD137])
* Has received prior radiotherapy to the thorax, including radiotherapy to the esophagus, mediastinum, or breast
* Has received a live vaccine within 30 days prior to the first dose of study intervention
* Has received an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention administration
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study treatment
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. A prior NSCLC that occurred and was treated curatively at least 2 years prior to the date of the current diagnosis would be considered a separate primary lung cancer, and therefore an additional malignancy. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast c carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Has a known hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has a known history of Hepatitis B or known active Hepatitis C virus infection
* Has an active autoimmune disease that has required systemic treatment in past 2 years, except replacement therapy
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of active tuberculosis (TB; Bacillus tuberculosis)
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of pembrolizumab/placebo and 180 days after the last radiotherapy dose
* Have not adequately recovered from major surgery or have ongoing surgical complications
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2025-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (194):
- United States (42):
  - University of Alabama ( Site 0099), Birmingham, Alabama
  - Infirmary Cancer Care ( Site 3044), Mobile, Alabama
  - Alaska Oncology and Hematology ( Site 3063), Anchorage, Alaska
  - Banner MD Anderson Cancer Center ( Site 3029), Gilbert, Arizona
  - CARTI Cancer Center ( Site 3045), Little Rock, Arkansas
  - USC Norris Comprehensive Cancer Center ( Site 0007), Los Angeles, California
  - Veterans Affairs Palo Alto Health Care System ( Site 3039), Palo Alto, California
  - National Jewish Health ( Site 0010), Denver, Colorado
  - Yale University ( Site 0011), New Haven, Connecticut
  - Mid Florida Hematology and Oncology Center ( Site 0067), Orange City, Florida
  - H. Lee Moffitt Cancer Center and Research Institute ( Site 0016), Tampa, Florida
  - Goshen Center for Cancer Care ( Site 0022), Goshen, Indiana
  - Franciscan Health Indianapolis ( Site 0024), Indianapolis, Indiana
  - University of Kentucky School of Medicine & Hospitals ( Site 0026), Lexington, Kentucky
  - Sinai Hospital of Baltimore ( Site 3011), Baltimore, Maryland
  - William E. Kahlert Regional Cancer Center ( Site 3031), Westminster, Maryland
  - Massachusetts General Hospital-Cancer Center Protocol Office ( Site 3007), Boston, Massachusetts
  - Mass General / North Shore Center for Outpatient Care ( Site 3040), Danvers, Massachusetts
  - University of Massachusetts ( Site 0029), Worcester, Massachusetts
  - Sanford Bemidji ( Site 0080), Bemidji, Minnesota
  - University of Minnesota ( Site 0069), Minneapolis, Minnesota
  - University of Missouri Hospital ( Site 3058), Columbia, Missouri
  - Cox Medical Center North-Cox Medical Center/Hulston Cancer Center/ Radiation Oncology ( Site 3060), Springfield, Missouri
  - St. Vincent Healthcare Frontier Cancer Center ( Site 3012), Billings, Montana
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 3036), Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey ( Site 0043), New Brunswick, New Jersey
  - Hematology-Oncology Associates of CNY ( Site 3055), East Syracuse, New York
  - Mount Sinai Hospital ( Site 0046), New York, New York
  - Westchester Medical Center ( Site 3057), Valhalla, New York
  - White Plains Hospital ( Site 3014), White Plains, New York
  - Sanford Health Roger Maris Cancer Center ( Site 0079), Fargo, North Dakota
  - Lehigh Valley Hospital- Cedar Crest ( Site 3005), Allentown, Pennsylvania
  - St. Luke's University Health Network ( Site 3006), Bethlehem, Pennsylvania
  - Penn State University Milton S. Hershey Medical Center ( Site 0064), Hershey, Pennsylvania
  - Fox Chase Cancer Center ( Site 0051), Philadelphia, Pennsylvania
  - Allegheny General Hospital ( Site 3028), Pittsburgh, Pennsylvania
  - Lankenau Medical Center ( Site 3041), Wynnewood, Pennsylvania
  - Sanford Cancer Center Oncology Clinic ( Site 0053), Sioux Falls, South Dakota
  - Mountain States Health Alliance ( Site 3054), Johnson City, Tennessee
  - University of Tennessee Medical Center Knoxville ( Site 3010), Knoxville, Tennessee
  - Vanderbilt University Medical Center ( Site 0075), Nashville, Tennessee
  - Cancer Care Northwest ( Site 0063), Spokane Valley, Washington
- Argentina (8):
  - Hospital Italiano de Buenos Aires-Clinical Oncology ( Site 0206), ABB, Buenos Aires F.D.
  - Hospital Britanico de Buenos Aires ( Site 0204), Buenos Aires, Buenos Aires F.D.
  - Sanatorio Parque ( Site 0207), Rosario, Santa Fe Province
  - Hospital Provincial del Centenario ( Site 0205), Rosario, Santa Fe Province
  - IDIM Instituto de Diagnostico e Investigaciones Metabolicas ( Site 0208), Buenos Aires
  - Hospital Aleman ( Site 0200), Buenos Aires
  - Instituto Medico Especializado Alexander Fleming ( Site 0203), Buenos Aires
  - CEMIC ( Site 0201), Buenos Aires
- Australia (5):
  - Port Macquarie Base Hospital ( Site 2500), Port Macquarie, New South Wales
  - GenesisCare North Shore ( Site 2508), St Leonards, New South Wales
  - Royal Brisbane and Women s Hospital ( Site 2502), Herston, Queensland
  - Icon Cancer Centre Hobart ( Site 2507), Hobart, Tasmania
  - Austin Health ( Site 2501), Melbourne, Victoria
- Austria (4):
  - Landeskrankenhaus - Universitatsklinikum Graz ( Site 0804), Graz, Styria
  - Universitatsklinik LKH Innsbruck ( Site 0802), Innsbruck, Tyrol
  - Keppler Universitatsklinikum ( Site 0806), Linz, Upper Austria
  - Social Medical Center - Otto Wagner Hospital ( Site 0801), Vienna, Vienna
- Brazil (8):
  - Irmandade da Santa Casa de Misericordia de Porto Alegre ( Site 0318), Porto Alegre, Rio Grande do Sul
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da Pucrs ( Site 0301), Porto Alegre, Rio Grande do Sul
  - Clínica de Oncologia Reichow ( Site 0319), Blumenau, Santa Catarina
  - Hospital e Maternidade Celso Pierro ( Site 0313), Campinas, São Paulo
  - Instituto Nacional Do Cancer Jose Alencar Gomes Da Silva ( Site 0305), Rio de Janeiro
  - Instituto do Cancer do Estado de Sao Paulo - ICESP ( Site 0300), São Paulo
  - Hospital Paulistano - Amil Clinical Research ( Site 0316), São Paulo
  - A.C. Camargo Cancer Center ( Site 0312), São Paulo
- Canada (9):
  - Moncton Hospital - Horizon Health Network ( Site 0105), Moncton, New Brunswick
  - Health Sciences North Research Institute ( Site 0107), Greater Sudbury, Ontario
  - Kingston Health Sciences Centre ( Site 0100), Kingston, Ontario
  - Trillium Health Partners - Credit Valley Hospital ( Site 0102), Mississauga, Ontario
  - The Ottawa Hospital ( Site 0104), Ottawa, Ontario
  - Sault Area Hospital ( Site 0101), Sault Ste. Marie, Ontario
  - CIUSSS de l Est de L Ile de Montreal - Hopital Maisonneuve-Rosemont ( Site 0110), Montreal, Quebec
  - McGill University Health Centre ( Site 0113), Montreal, Quebec
  - CHUS - Hopital Fleurimont ( Site 0111), Sherbrooke, Quebec
- France (9):
  - CHU Poitiers ( Site 1109), Poitiers, Ain
  - CHU de Brest -Site Hopital Morvan ( Site 1100), Brest, Finistere
  - Institut Bergonie ( Site 1102), Bordeaux, Gironde
  - Institut Regional du Cancer de Montpellier - ICM ( Site 1108), Montpellier, Herault
  - CHU de Rouen ( Site 1113), Rouen, Seine-Maritime
  - Hopital Sud du Amiens ( Site 1115), Amiens, Somme
  - Institut Curie ( Site 1112), Paris
  - Hopital Cochin ( Site 1107), Paris
  - A.P.H. Paris. Hopital Bichat Claude Bernard ( Site 1114), Paris
- Germany (8):
  - Klinikum Esslingen-Klinik für Kardiologie und Pneumologie ( Site 1208), Esslingen am Neckar, Baden-Wurttemberg
  - Universitaetsklinikum Heidelberg. ( Site 1204), Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen ( Site 1209), Erlangen, Bavaria
  - UKGM Gießen/Marburg-Medical Clinic V ( Site 1210), Giessen, Hesse
  - Pius Hospital Oldenburg ( Site 1202), Oldenburg, Lower Saxony
  - Universitaetsklinikum Essen ( Site 1201), Essen, North Rhine-Westphalia
  - Evangelisches Krankenhaus Hamm gGmbH ( Site 1205), Hamm, North Rhine-Westphalia
  - Charite Universitaetsmedizin Berlin ( Site 1207), Berlin
- Hungary (14):
  - Pécsi Tudományegyetem Klinikai Központ-Onkoterápiás Intézet ( Site 2314), Pécs, Baranya
  - CRU Hungary KFT ( Site 2309), Miskolc, Borsod-Abauj Zemplen county
  - Bacs-Kiskun Varmegyei Oktatokorhaz-Onkoradiologiai Kozpont ( Site 2311), Kecskemét, Bács-Kiskun county
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz ( Site 2312), Székesfehérvár, Fejér
  - Petz Aladar Megyei Oktato Korhaz ( Site 2305), Győr, Győr-Moson-Sopron
  - Debreceni Egyetem Klinikai Kozpont ( Site 2301), Debrecen, Hajdú-Bihar
  - Jász-Nagykun-Szolnok Vármegyei Hetényi Géza Kórház ( Site 2310), Szolnok, Jász-Nagykun-Szolnok
  - Törökbálinti Tüdőgyógyintézet ( Site 2302), Törökbálint, Pest County
  - Somogy Megyei Kaposi Mor Oktato Korhaz ( Site 2307), Kaposvár, Somogy County
  - Farkasgyepui Tudogyogyintezet ( Site 2313), Farkasgyepű, Veszprém megye
  - Semmelweis University ( Site 2303), Budapest
  - Orszagos Koranyi Pulmonologiai Intezet ( Site 2304), Budapest
  - Orszagos Koranyi Pulmonologiai Intezet ( Site 2306), Budapest
  - Orszagos Onkologiai Intezet ( Site 2308), Budapest
- Italy (5):
  - Ospedale Santissima Annunziata ( Site 1303), Chieti
  - A.O. Universitaria Careggi ( Site 1301), Florence
  - Policlinico di Modena ( Site 1306), Modena
  - Policlinico Agostino Gemelli ( Site 1302), Roma
  - Azienda Ospedaliera S. Giovanni Addolorata-Oncologia Medica ( Site 1309), Roma
- Japan (17):
  - Aichi Cancer Center Hospital ( Site 2804), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 2800), Kashiwa, Chiba
  - Kurume University Hospital ( Site 2815), Kurume, Fukuoka
  - Kobe Minimally Invasive Cancer Center ( Site 2811), Kobe, Hyōgo
  - University of Tsukuba Hospital ( Site 2809), Tsukuba, Ibaraki
  - Sendai Kousei Hospital ( Site 2814), Sendai, Miyagi
  - Kansai Medical University Hospital ( Site 2808), Hirakata, Osaka
  - Osaka Medical and Pharmaceutical University Hospital ( Site 2813), Takatsuki, Osaka
  - University of Yamanashi Hospital ( Site 2807), Chūō, Yamanashi
  - Chiba University Hospital ( Site 2806), Chiba
  - National Hospital Organization Kyushu Cancer Center ( Site 2816), Fukuoka
  - Hiroshima University Hospital ( Site 2810), Hiroshima
  - Niigata Cancer Center Hospital ( Site 2801), Niigata
  - Osaka International Cancer Institute ( Site 2812), Osaka
  - Tokyo Metropolitan Komagome Hospital ( Site 2802), Tokyo
  - The Cancer Institute Hospital of JFCR ( Site 2803), Tokyo
  - Showa University Hospital ( Site 2805), Tokyo
- Netherlands (3):
  - Ziekenhuis Rijnstate ( Site 1405), Arnhem, Gelderland
  - Tergooiziekenhuizen, locatie Hilversum-Oncology ( Site 1407), Hilversum, North Holland
  - Meander Medisch Centrum-Studie Team Oncologie ( Site 1403), Amersfoort, Utrecht
- Auckland City Hospital ( Site 2900), Grafton, Auckland, New Zealand
- Norway (3):
  - St Olavs Hospital ( Site 1504), Trondheim, Sor-Trondelag
  - Helse Bergen HF Haukeland Universitetssykehus ( Site 1502), Bergen, Vestfold
  - Oslo Universitetssykehus HF Ulleval Sykehus ( Site 1500), Oslo
- Poland (6):
  - Centrum Onkologii im. prof. Franciszka ukaszczyka-Ambulatorium Chemioterapii ( Site 2407), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie ( Site 2400), Krakow, Lesser Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie (, Warsaw, Masovian Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach ( Site 2403), Gliwice, Silesian Voivodeship
  - SPZOZ MSWIA z Warminsko-Mazurskim Centrum Onkologii w Olsztynie ( Site 2404), Olsztyn, Warmian-Masurian Voivodeship
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii ( Site 2402), Lodz, Łódź Voivodeship
- Romania (2):
  - Amethyst Radiotherapy Center-Oncologie Medicala ( Site 3201), Florești, Cluj
  - Institutul Oncologic-Oncologie Medicala ( Site 3202), Cluj-Napoca
- Russia (8):
  - Chelyabinsk Regional Clinical Oncology Dispensary ( Site 2014), Chelyabinsk, Chelyabinsk Oblast
  - GUZ Lipetsk Regional Oncology Dispensary ( Site 2010), Lipetsk, Lipetsk Oblast
  - N.N.Blokhin Russian Cancer Research center ( Site 2013), Moscow, Moscow
  - Russian Scientific Center of Roentgenoradiology ( Site 2011), Moscow, Moscow
  - Medical institute named after Berezin Sergey ( Site 2009), Saint Petersburg, Sankt-Peterburg
  - Scientific Research Oncology Institute n.a. N.N.Petrov ( Site 2000), Saint Petersburg, Sankt-Peterburg
  - Sverdlovsk Regional Oncology Hospital ( Site 2012), Yekaterinburg, Sverdlovsk Oblast
  - Republican Clinical Oncology Dispensary of Tatarstan MoH ( Site 2001), Kazan', Tatarstan, Respublika
- South Korea (5):
  - National Cancer Center ( Site 2604), Goyang-si, Kyonggi-do
  - The Catholic University of Korea St. Vincent s Hospital ( Site 2606), Gyeonggi-do, Kyonggi-do
  - Chungbuk National University Hospital ( Site 2605), Cheongju-si, North Chungcheong
  - Seoul National University Hospital ( Site 2600), Seoul
  - Samsung Medical Center ( Site 2603), Seoul
- Spain (4):
  - Hospital Universitario Quiron Madrid ( Site 1601), Pozuelo de Alarcón, Madrid
  - Hospital Universitario La Fe ( Site 1603), Valencia, Valenciana, Comunitat
  - Hospital General Universitari Vall d Hebron ( Site 1602), Barcelona
  - Hospital General Universitario Gregorio Maranon ( Site 1604), Madrid
- Switzerland (2):
  - Hopitaux Universitaires de Geneve HUG ( Site 1706), Geneva, Canton of Geneva
  - Universitaetsspital Zuerich ( Site 1700), Zurich, Canton of Zurich
- Taiwan (4):
  - Tri-Service General Hospital ( Site 3300), Taipei City, Taipei
  - Kaohsiung Medical University Chung-Ho Memorial Hospital ( Site 3304), Kaohsiung City
  - Taipei Medical University Hospital ( Site 3303), Taipei
  - Taipei Veterans General Hospital ( Site 3301), Taipei
- Turkey (Türkiye) (8):
  - Baskent Adana Dr Turgut Noyan Uygulama ve Arastirma Merkezi ( Site 2105), Adana
  - Hacettepe University Medical Faculty ( Site 2100), Ankara
  - Dr Abdurrahman Yurtaslan Oncology Training and Research Hospital ( Site 2101), Ankara
  - Göztepe Prof. Dr. Süleyman Yalçın Şehir Hastanesi-oncology ( Site 2116), Istanbul
  - Kartal Training and Research Hospital ( Site 2102), Istanbul
  - I.E.U. Medical Point Hastanesi ( Site 2115), Izmir
  - Erciyes University Medical Faculty ( Site 2109), Kayseri
  - Sakarya Universitesi Tip Fakultesi Hastanesi ( Site 2114), Sakarya
- Ukraine (7):
  - Medical center Medikal Plaza of Ecodnipro LLC ( Site 2207), Dnipro, Dnipropetrovsk Oblast
  - Regional Centre of Oncology-Thoracic organs ( Site 2202), Kharkiv, Kharkivs’ka Oblast’
  - Ukrainian Center of Tomotherapy ( Site 2206), Kropyvnitskiy, Kirovohrad Oblast
  - Medical Center of Yuriy Spizhenko LLC.-Clinical Trial ( Site 2205), Kapitanivka Village, Kyivska Oblast
  - Medical Center Asklepion LLC ( Site 2208), Khodosovka, Kyivska Oblast
  - Medical and Diagnostic Centre LLC Dobryi Prognoz ( Site 2203), Kyiv, Kyivska Oblast
  - Kyiv City Clinical Oncology Centre ( Site 2200), Kyiv
- United Kingdom (12):
  - University Hospitals Bristol NHS Foundation Trust ( Site 1802), Bristol, Bristol, City of
  - Royal Free London NHS Foundation Trust ( Site 1813), London, Camden
  - Weston Park Hospital ( Site 1801), Sheffield, Derbyshire
  - Clatterbridge Cancer Center NHS FT ( Site 1800), Liverpool, England
  - Lancashire Teaching Hospitals NHS Foundation Trust ( Site 1809), Preston, Lancashire
  - Leicester Royal Infirmary ( Site 1811), Leicester, Leicestershire
  - University College London Hospital NHS Foundation Trust ( Site 1806), London, London, City of
  - Guy s and St Thomas Hospital NHS Foundation Trust ( Site 1808), London, London, City of
  - Norfolk and Norwich University Foundation NHS Trust ( Site 1805), Norwich, Norfolk
  - Oxford University Hospitals NHS Foundation Trust ( Site 1812), Oxford, Oxfordshire
  - Darlington Memorial Hospital NHS Trust ( Site 1810), Darlington
  - Mount Vernon Hospital ( Site 1803), Northwood

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Swaminath A, Parpia S, Wierzbicki M, Kundapur V, Faria S, Okawara GS, Tsakiridis TK, Ahmed N, Bujold A, Hirmiz K, Owen T, Leong N, Ramchandar K, Filion E, Lau H, Gabos Z, Thompson R, Yaremko B, Mehiri S, Louie AV, Quan K, Levine MN, Wright JR, Whelan TJ. Stereotactic vs Hypofractionated Radiotherapy for Inoperable Stage I Non-Small Cell Lung Cancer: The LUSTRE Phase 3 Randomized Clinical Trial. JAMA Oncol. 2024 Nov;10(11):1571-1575. doi: 10.1001/jamaoncol.2024.3089. Epub 2024 Sep 19. PMID 39298144
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26213&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female participants at least 18 years of age with unresected Stage I or II (limited Stage IIB N0, M0) Non-Small Cell Lung Cancer (NSCLC) who had received no prior anticancer therapy for their present lung cancer were recruited.
Pre-assignment Details: Of 737 participants screened, 448 were randomized 1:1 to receive either stereotactic body radiotherapy (SBRT) plus pembrolizumab or SBRT plus placebo.
Groups:
- SBRT + Pembrolizumab: Participants received SBRT once every 3 days for 3, 4, 5, or 8 fractions (dependent on tumor type/location; 45-70 Gray [Gy] total) over approximately 2 weeks PLUS pembrolizumab 200 mg via IV infusion once every 3 weeks for up to 17 cycles (up to approximately 1 year). Each cycle was 21 days.
- SBRT + Placebo: Participants received SBRT once every 3 days for 3, 4, 5, or 8 fractions (dependent on tumor type/location; 45-70 Gy total) over approximately 2 weeks PLUS placebo (normal saline solution) via IV infusion once every 3 weeks for up to 17 cycles (up to approximately 1 year). Each cycle was 21 days.
Period: Overall Study
Arm/Group | SBRT + Pembrolizumab | SBRT + Placebo
Started | 227 | 221
Treated | 226 | 218
Completed | 0 | 0
Not Completed | 227 | 221
Not completed — Death | 73 | 62
Not completed — Lost to Follow-up | 3 | 0
Not completed — Physician Decision | 0 | 3
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Study Terminated By Sponsor | 144 | 153

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SBRT + Pembrolizumab | SBRT + Placebo | Total
Number analyzed (Participants) | 227 | 221 | 448
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.2 (8.0) | 72.4 (7.6) | 72.8 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 100 | 189
  Male | 138 | 121 | 259
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 20 | 43
  Not Hispanic or Latino | 190 | 186 | 376
  Unknown or Not Reported | 14 | 15 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 31 | 26 | 57
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 183 | 177 | 360
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 9 | 9 | 18
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) Score [Count of Participants; unit: Participants] — The ECOG PS Score describes a participant's level of functioning in terms of their ability to care for themself, daily activity, and physical ability, and ranges from 0 (fully active) to 5 (dead). An ECOG PS of 0 (Fully active, able to carry on all pre-disease performance without restriction), 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature), or 2 (Ambulatory and capable of all self-care, but unable to carry out any work activities) was required for inclusion in the study and used to stratify randomization.
  Participants
    ECOG PS 0 = Normal activity | 86 | 84 | 170
    ECOG PS 1 = Symptoms, but ambulatory | 122 | 122 | 244
    ECOG PS 2 = Ambulatory, capable of selfcare, unable to carry out work activities | 19 | 15 | 34
NSCLC Disease Stage [Count of Participants; unit: Participants] — Participants were categorized as NSCLC Stage I or NSCLC Stage II according to the American Joint Committee on Cancer Manual 8th Edition (AJCC V8). NSCLC stages range from I to IV, with higher stage numbers indicating that the cancer is more advanced. NSCLC Stage (I or II) was used as a randomization stratification factor.
  Participants
    Stage I | 204 | 197 | 401
    Stage II | 23 | 24 | 47
Geographic Region of Enrollment Site [Count of Participants; unit: Participants] — Geographic region of enrolment site (East Asia versus non-East Asia) was used as a randomization stratification factor.
  Participants
    East Asia | 29 | 26 | 55
    Non-East Asia | 198 | 195 | 393
Reason for not Receiving Surgery [Count of Participants; unit: Participants] — The "Reason for not receiving surgery" (medically inoperable versus refused surgery) was used as a randomization stratification factor.
  Participants
    Refused Surgery | 43 | 36 | 79
    Medically Inoperable | 184 | 185 | 369

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS)
Description: EFS was defined as the time from randomization to the first occurrence of any of the following events: 1) local, regional, or distant recurrence of disease as assessed by radiographic recurrence by blinded independent central review (BICR), positive pathology by local assessment, physical examination by local assessment confirmed by positive pathology and/or radiographic recurrence by BICR, OR 2) death due to any cause. EFS was reported for each arm.
Time Frame: Up to approximately 56.8 months
Population: All randomized participants were analyzed according to the treatment arm they were randomized to.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SBRT + Pembrolizumab | SBRT + Placebo
Number analyzed (Participants) | 227 | 221
months | 31.2 [22.5 to 39.1] | 28.3 [19.8 to 33.1]
Statistical Analysis 1: Comparison: SBRT + Pembrolizumab vs SBRT + Placebo; Hazard ratio and 95% confidence intervals (CIs) were based on Cox regression model with Efron's method of tie handling with treatment as a covariate, stratified by Disease Stage (Stage I versus Stage II), ECOG Performance Status (0 or 1 versus 2), Geographic Region of Enrollment Site (East Asia versus non-East Asia), and Reason For Not Receiving Surgery ("medically inoperable" versus "refused surgery"); Test type: Superiority; p = 0.29320, Log Rank — 1-sided p-value based on log-rank test stratified by Disease Stage, ECOG Performance Status, Geographic Region of Enrollment Site, and Reason For Not Receiving Surgery; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.69 to 1.24]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date of randomization to date of death from any cause. OS was reported for each arm.
Time Frame: Up to approximately 56.8 months
Population: All randomized participants were analyzed according to the treatment arm they were randomized to.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SBRT + Pembrolizumab | SBRT + Placebo
Number analyzed (Participants) | 227 | 221
months | 54.7 [33.5 to NA] — NA = Kaplan-Meier estimate for OS upper 95% confidence limit was not reached at time of data cut-off due to an insufficient number of participants with an event. | NA [44.4 to NA] — NA = Kaplan-Meier estimates for median OS and OS upper 95% confidence limit were not reached at time of data cut-off due to an insufficient number of participants with an event.
Statistical Analysis 1: Comparison: SBRT + Pembrolizumab vs SBRT + Placebo; Hazard ratio and 95% CIs were based on Cox regression model with Efron's method of tie handling with treatment as a covariate, stratified by Disease Stage (Stage I versus Stage II), ECOG Performance Status (0 or 1 versus 2), Geographic Region of Enrollment Site (East Asia versus non-East Asia), and Reason for Not Receiving Surgery ("medically inoperable" versus "refused surgery"); Test type: Other; p = 0.93971, Log Rank — [p-value comment as in outcome 1, analysis 1]; Per protocol, since the EFS null hypothesis was not rejected, the OS hypothesis was not formally tested and the p-value should be considered nominal; Hazard Ratio (HR) = 1.33, 95% CI 2-sided [0.93 to 1.90]

3. Secondary Outcome: Time to Death or Distant Metastases (TDDM)
Description: TTDM was defined as the time from randomization to the first documented distant metastases or death from any cause, whichever occurred first. The TDDM was reported for each arm.
Time Frame: Up to approximately 56.8 months
Population: All randomized participants were analyzed according to the treatment arm they were randomized to.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SBRT + Pembrolizumab | SBRT + Placebo
Number analyzed (Participants) | 227 | 221
months | 39.1 [30.5 to NA] — NA = Kaplan-Meier estimate for TDDM upper 95% confidence limit was not reached at time of data cut-off due to an insufficient number of participants with an event. | 41.3 [31.1 to NA] — NA = Kaplan-Meier estimate for TDDM upper 95% confidence limit was not reached at time of data cut-off due to an insufficient number of participants with an event.
Statistical Analysis 1: Comparison: SBRT + Pembrolizumab vs SBRT + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; Per protocol, there was no hypothesis pre-specified for TDDM to be formally tested; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.74 to 1.42]

4. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experienced an AE were reported.
Time Frame: Up to approximately 64 months
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT + Pembrolizumab | SBRT + Placebo
Number analyzed (Participants) | 226 | 218
Participants | 217 | 200

5. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinued study treatment due to an AE were reported.
Time Frame: Up to approximately 16 months
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT + Pembrolizumab | SBRT + Placebo
Number analyzed (Participants) | 226 | 218
Participants | 62 | 25

6. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status/Quality of Life (Items 29 and 30) Score
Description: The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" were scored on a 7-point scale (1=Very Poor to 7=Excellent). The combined score of Global Health Status (EORTC QLQ-C30 Item 29) and Quality of Life (EORTC QLQ-C30 Item 30) was computed by averaging the raw scores of the 2 items and then applying a linear transformation to standardize the average score, so that the combined scores ranged from 0-100. A higher score indicates a better outcome. The change from baseline in GHS/QoL combined score was reported for each arm.
Time Frame: Baseline and up to 24 weeks
Population: All randomized participants who received at least 1 dose of study intervention and had at least 1 EORTC QLQ-C30 assessment available were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | SBRT + Pembrolizumab | SBRT + Placebo
Number analyzed (Participants) | 225 | 214
Score on a Scale | -2.17 [-5.00 to 0.66] | -0.96 [-3.78 to 1.86]
Statistical Analysis 1: Comparison: SBRT + Pembrolizumab vs SBRT + Placebo; Stats: LS Mean change and 95% CIs were based on a constrained longitudinal data analysis (cLDA) model with the EORTC QLQ-C30 scores as the response variable with covariates for treatment by study visit interaction, and stratification factors by Disease Stage (Stage I versus Stage II), ECOG Performance Status (0 or 1 versus 2), Geographic Region of Enrollment Site (East Asia versus non-East Asia), and Reason For Not Receiving Surgery (medically inoperable versus refused surgery); Test type: Other; p = 0.5187, cLDA model; Mean Difference (Final Values) = -1.21, 95% CI 2-sided [-4.90 to 2.48]

7. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer Module 13 (EORTC QLQ-LC13) Cough (Item 31) Score
Description: The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant responses to the EORTC QLQ-LC13 question "How much did you cough?" were scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores were standardized, so that scores ranged from 0 to 100. A lower score indicates a better outcome. The change from baseline in cough (EORTC QLQ LC13 Item 31) score was reported for each arm.
Time Frame: Baseline and up to 24 weeks
Population: All randomized participants who received at least 1 dose of study intervention and had at least 1 EORTC QLQ-LC13 assessment available were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | SBRT + Pembrolizumab | SBRT + Placebo
Number analyzed (Participants) | 225 | 214
Score on a scale | -1.44 [-5.23 to 2.36] | 2.91 [-0.87 to 6.68]
Statistical Analysis 1: Comparison: SBRT + Pembrolizumab vs SBRT + Placebo; LS Mean change and 95% CIs were based on a cLDA model with the EORTC QLQ-LC13 scores as the response variable with covariates for treatment by study visit interaction, and stratification factors by Disease Stage (Stage I versus Stage II), ECOG Performance Status (0 or 1 versus 2), Geographic Region of Enrollment Site (East Asia versus non-East Asia), and Reason For Not Receiving Surgery (medically inoperable versus refused surgery); Test type: Other; p = 0.0906, cLDA model; Mean Difference (Final Values) = -4.34, 95% CI 2-sided [-9.38 to 0.69]

8. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer Module 13 (EORTC QLQ-LC13) Chest Pain (Item 40) Score
Description: The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant responses to the question "Have you had pain in your chest?" were scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores were standardized, so that scores ranged from 0 to 100. A lower score indicates a better outcome. The change from baseline in chest pain (EORTC QLQ-LC13 Item 40) score was reported for each arm.
Time Frame: Baseline and up to 24 weeks
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | SBRT + Pembrolizumab | SBRT + Placebo
Number analyzed (Participants) | 225 | 214
Score on a Scale | 3.00 [-0.09 to 6.10] | 1.76 [-1.32 to 4.84]
Statistical Analysis 1: Comparison: SBRT + Pembrolizumab vs SBRT + Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.5482, cLDA model; Mean Difference (Final Values) = 1.24, 95% CI 2-sided [-2.83 to 5.31]

9. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Dyspnea (Item 8) Score
Description: The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the question "Were you short of breath?" were scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores were standardized, so that scores ranged from 0 to 100. A lower score indicates a better outcome. The change from baseline in dyspnea (EORTC QLQ-C30 Item 8) score was reported for each arm.
Time Frame: Baseline and up to 24 weeks
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | SBRT + Pembrolizumab | SBRT + Placebo
Number analyzed (Participants) | 225 | 214
Score on a Scale | -1.80 [-5.95 to 2.36] | -0.81 [-4.94 to 3.32]
Statistical Analysis 1: Comparison: SBRT + Pembrolizumab vs SBRT + Placebo; LS Mean change and 95% CIs were based on a cLDA model with the EORTC QLQ-C30 scores as the response variable with covariates for treatment by study visit interaction, and stratification factors by Disease Stage (Stage I versus Stage II), ECOG Performance Status (0 or 1 versus 2), Geographic Region of Enrollment Site (East Asia versus non-East Asia), and Reason For Not Receiving Surgery (medically inoperable versus refused surgery); Test type: Other; p = 0.7253, cLDA model; Mean Difference (Final Values) = -0.99, 95% CI 2-sided [-6.50 to 4.53]

10. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30) Physical Functioning (Items 1-5) Score
Description: The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to 5 questions about their physical functioning were scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores were standardized, so that scores ranged from 0 to 100. A higher score indicates a better quality of life. The change from baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) combined score was reported for each arm.
Time Frame: Baseline and up to 24 weeks
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | SBRT + Pembrolizumab | SBRT + Placebo
Number analyzed (Participants) | 225 | 214
Score on a Scale | -0.52 [-3.08 to 2.03] | -0.31 [-2.86 to 2.24]
Statistical Analysis 1: Comparison: SBRT + Pembrolizumab vs SBRT + Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Other; p = 0.9055, cLDA model; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-3.70 to 3.28]

ADVERSE EVENTS:
Time Frame: Up to approximately 64 months
Description: All-Cause Mortality reported for all randomized participants.
  Serious AEs and Other AEs were reported for all randomized participants who received at least 1 dose of study treatment. Per protocol, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug were excluded as AEs.
Groups:
- Pembrolizumab + SBRT: Participants received SBRT once every 3 days for 3, 4, 5, or 8 fractions (dependent on tumor type/location; 45-70 Gray [Gy] total) over approximately 2 weeks PLUS pembrolizumab 200 mg via IV infusion once every 3 weeks for up to 17 cycles (up to approximately 1 year). Each cycle was 21 days.
- Placebo + SBRT: Participants received SBRT once every 3 days for 3, 4, 5, or 8 fractions (dependent on tumor type/location; 45-70 Gy total) over approximately 2 weeks PLUS placebo (normal saline solution) via IV infusion once every 3 weeks for up to 17 cycles (up to approximately 1 year). Each cycle was 21 days.
Arm/Group | Pembrolizumab + SBRT | Placebo + SBRT
All-Cause Mortality (participants affected / at risk) | 76/227 | 63/221
Serious Adverse Events (participants affected / at risk) | 90/226 | 74/218
Other Adverse Events (participants affected / at risk) | 198/226 | 176/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + SBRT (N=226) | Placebo + SBRT (N=218)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Aplasia pure red cell (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 3 (3) | 2 (3)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Dilated cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Immune-mediated hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 0 (0)
Drowning (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0)
Abscess oral (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 5 (5)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 6 (6)
Catheter site infection (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 19 (23) | 7 (7)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 6 (6) | 2 (2)
Prostate infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (7) | 0 (0)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (4) | 2 (3)
Encephalitis autoimmune (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 16 (24) | 10 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + SBRT (N=226) | Placebo + SBRT (N=218)
Anaemia (Blood and lymphatic system disorders) | 28 (32) | 15 (18)
Hyperthyroidism (Endocrine disorders) | 13 (13) | 5 (5)
Hypothyroidism (Endocrine disorders) | 37 (41) | 10 (10)
Constipation (Gastrointestinal disorders) | 20 (23) | 21 (23)
Diarrhoea (Gastrointestinal disorders) | 38 (52) | 31 (43)
Nausea (Gastrointestinal disorders) | 17 (22) | 25 (30)
Vomiting (Gastrointestinal disorders) | 18 (20) | 8 (11)
Asthenia (General disorders) | 20 (22) | 18 (22)
Chest pain (General disorders) | 15 (18) | 16 (22)
Fatigue (General disorders) | 51 (61) | 43 (48)
Oedema peripheral (General disorders) | 12 (12) | 15 (17)
Pyrexia (General disorders) | 14 (17) | 5 (5)
COVID-19 (Infections and infestations) | 12 (12) | 16 (18)
Pneumonia (Infections and infestations) | 12 (14) | 10 (12)
Urinary tract infection (Infections and infestations) | 11 (16) | 16 (20)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 20 (22) | 19 (20)
Alanine aminotransferase increased (Investigations) | 17 (23) | 10 (12)
Aspartate aminotransferase increased (Investigations) | 15 (18) | 10 (11)
Blood creatinine increased (Investigations) | 20 (28) | 20 (25)
Decreased appetite (Metabolism and nutrition disorders) | 26 (27) | 16 (16)
Hyperglycaemia (Metabolism and nutrition disorders) | 18 (24) | 8 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 12 (13) | 8 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 40 (49) | 16 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (17) | 18 (19)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (17) | 13 (14)
Dizziness (Nervous system disorders) | 14 (14) | 13 (14)
Headache (Nervous system disorders) | 13 (15) | 19 (22)
Insomnia (Psychiatric disorders) | 16 (16) | 13 (13)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 16 (20) | 10 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 34 (39) | 39 (46)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 41 (47) | 39 (42)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 15 (19) | 7 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 10 (10) | 13 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 39 (44) | 21 (35)
Rash (Skin and subcutaneous tissue disorders) | 36 (53) | 16 (20)
Hypertension (Vascular disorders) | 13 (15) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will comply with the requirements for publication of study results, and will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT03924869/Prot_SAP_000.pdf